CLINICAL TRIAL: NCT05317884
Title: Evaluation of Email-based Reminders in Promoting Adherence to the Recommended Pediatric Preventative-visit Schedule Among Rural Patients
Brief Title: Email-based Reminders Promoting Recommended Pediatric Preventative Visits
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Geisinger Clinic (Other)
Responsible Party: Principal Investigator, Amir Goren, Program Director, Behavioral Insights Team, Geisinger Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2021-0106
Record Dates: First submitted 2022-03-22; First posted 2022-04-08 (Actual); Last update posted 2022-11-23 (Actual); Status verified 2022-11

CONDITIONS: Immunization Programs
Keywords: Pediatrics; Reminder Systems; Preventive Medicine; Child Health; Appointments and Schedules

STUDY DESIGN:
Intervention Model Description: No reminder group vs. reminder group
Who Masked: Participant, Care Provider
Masking Description: The participants and providers will not know that email reminders were randomized. Participants who received an email (and their providers if they shared this email) will know that they have received an email, but it is not likely that they will know that other participants did not receive an email (and vice-versa).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No Contact (No Intervention): No reminder sent
- Reminder (Experimental): Reminder email with contact information to set an appointment will be sent 12 weeks before the appointment.
  Interventions: Behavioral: Reminder

INTERVENTIONS:
Behavioral: Reminder — Email
  Arms: Reminder

SUMMARY:
The purpose of this study is to assess, prospectively, the effect of email reminders for well-child check (WCC) visits on adherence to these visits among those who have not yet scheduled the visit. The investigators hypothesize that sending reminders will increase scheduling WCC visits, attending WCC visits, and being up to date for the child's required immunizations beyond what occurs in the absence of these reminders.

DETAILED DESCRIPTION:
Regular attendance at recommended WCC visits is associated with having up-to-date immunizations. Standard care involves scheduling a follow-up WCC visit at the end of the current visit. However, if the child's parents do not choose to schedule a follow-up visit at that time or miss a WCC visit, they may not be offered another easy opportunity to schedule one. That is, they would have to remember to schedule a visit and contact the clinic proactively.

In this study, 30 days before a child is due for their WCC visit, parents who have not yet scheduled a WCC visit for up to 30 days (for 5-month-olds) or 60 days (for all other ages) after their child is due for a visit will be randomly assigned to two groups with a random number generator. One group will receive an email reminder, while the other group will not receive any reminder.

The randomization of participants to different conditions will be in place until 800 participants have been identified and randomly assigned to one of the arms (estimated sample to detect at least a 10% absolute difference) or 180 days, whichever comes first. To account for delays in updating clinical databases, the final outcome data will be checked 90 days after the last eligible visit (for a maximum study period of 270 days).

ELIGIBILITY:
Inclusion Criteria:

* Parents (or contact on record) of children aged 5, 8, 11, 14, or 17 months
* No WCC visits scheduled 30 days after the child's monthly birthday (for 5 month-olds) or 60 days (for all other ages) ahead of their due date for a WCC (i.e., month 6, 9, 12, 15, or 18)
* Has an email address on record
* Child is currently seen in Pediatric clinics under the Geisinger umbrella (has at least one prior visit)

Exclusion Criteria:

* Did not opt out of emails

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1186 (Actual)
Dates: Start 2022-05-16 (Actual); Primary Completion 2022-09-13 (Actual); Study Completion 2022-09-13 (Actual)

PRIMARY OUTCOMES:
WCC visit scheduled | 30-60 days from the email send date
  Binary variable of scheduling a WCC visit as established by visit type, visit reasons, and billing codes (if available)

SECONDARY OUTCOMES:
WCC visit made | 30-60 days from the email send date
  Binary variable of going to a WCC visit as established by billing codes
Immunization status | 60 days from the email send date
  Binary variable indicating whether pediatric vaccinations are up to date, defined as having no current immunization care gaps

OTHER OUTCOMES:
Emails opened | 60 days from the email send date
  Binary variable of opening the email
Follow-up WCC visit scheduled | 61-150 days from the email send date
  Binary variable of scheduling a WCC visit as established by visit type, visit reasons, and billing codes (if available)
Measles, Mumps, and Rubella immunization status | 60 days from the email send date
  Binary variable indicating whether Measles, Mumps, and Rubella (MMR) vaccinations are up to date, defined as having no current immunization care gaps
Hepatitis A immunization status | 60 days from the email send date
  Binary variable indicating whether Hepatitis A vaccinations are up to date, defined as having no current immunization care gaps
Hepatitis B immunization status | 60 days from the email send date
  Binary variable indicating whether Hepatitis B vaccinations are up to date, defined as having no current immunization care gaps
Varicella immunization status | 60 days from the email send date
  Binary variable indicating whether Varicella vaccinations are up to date, defined as having no current immunization care gaps

CONTACTS AND LOCATIONS:
Overall Officials: Amir Goren, PhD, Principal Investigator — Program Director, Behavioral Insights Team
Locations (1):
- Geisinger, Danville, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Data with no personally identifiable information will be made available to other researchers on the Open Science Framework for transparency. This will include the essential data and code needed to replicate the analysis that yielded reported findings. The PI did not examine or analyze any data from this study prior to this registration.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: The data will become available after publication of study results in a scientific journal and will be available as long as the Open Science Framework hosts the data.
Access Criteria: The data on the Open Science Framework will be open to anyone requesting that information.
URL: http://osf.io

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-08): https://cdn.clinicaltrials.gov/large-docs/84/NCT05317884/Prot_SAP_000.pdf